CLINICAL TRIAL: NCT04186026
Title: Effect of Combination of the Gut Hormones Neurotensin and GLP-1 on Physiological Regulation of Appetite and Food Intake
Brief Title: Co-infusion of Neurotensin and GLP-1 Effects on Appetite and Food Intake.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Birgitte Holst, Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 514-0386/19-3000
Record Dates: First submitted 2019-11-26; First posted 2019-12-04 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Obesity
Keywords: Neurotensin; Glucagon like peptide-1 (GLP-1)
MeSH Terms: conditions — Obesity | interventions — Sodium Chloride; Neurotensin; Glucagon-Like Peptide 1

STUDY DESIGN:
Intervention Model Description: Participants will be studied on multiple occasions (4 days) in a randomised and double blinded fashion.
Who Masked: Participant, Investigator
Masking Description: Participants will not be informed of the nature of the infusion they are administered on any of the study days. The investigator will be provided with an infusion (either isotonic saline with humane serum albumine (HSA) or isotonic saline with HSA + neurotensin or isotonic saline with HSA + GLP-1) prepared by a designated colleague
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Saline+Saline (Other)
  Interventions: Other: Saline + saline
- Neurotensin+Saline (Other)
  Interventions: Other: Neurotensin + saline
- GLP-1+Saline (Other)
  Interventions: Other: GLP-1 + saline
- Neurotensin + GLP-1 (Other)
  Interventions: Other: GLP-1 + Neurotensin

INTERVENTIONS:
Other: Saline + saline — Double saline infusion followed by an ad libitum meal
  Arms: Saline+Saline
Other: Neurotensin + saline — Neurotensin + saline infusion followed by an ad libitum meal
  Arms: Neurotensin+Saline
Other: GLP-1 + saline — GLP-1 + saline infusion followed by an ad libitum meal
  Arms: GLP-1+Saline
Other: GLP-1 + Neurotensin — GLP-1 + Neurotensin infusion followed by an ad libitum meal
  Arms: Neurotensin + GLP-1

SUMMARY:
Co-infusion of Neurotensin and GLP-1 Effects on Appetite and Food Intake.

DETAILED DESCRIPTION:
Neurotensin (NT), a gut hormone and neuropeptide, and GLP-1, as well a gut hormone, increases in circulation after bariatric surgery in rodents and humans and inhibit food intake in mice.

Studies in rodents have shown that a GLP-1 receptor agonist and long acting neurotensin inhibit food intake.

This study investigates whether the synergistic anorexic effects of neurotensin and GLP-1 agonism suggested by animal studies can be translated.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Above 18 years of age
* Normal hemoglobin concentration
* 28<BMI<40 kg/m2

Exclusion Criteria:

* Diabetes mellitus
* Truncal vagotomy
* Resection of intestine (apart from appendectomy)
* Tobaccos use
* Nephropathy (serum-creatinin>130 micromolar or/and albuminuria)
* Liver disease (Alanine transaminase or/and aspartate transaminase>2 times normal range.)
* Treatment with medication that cannot be paused in 12 hours
* Allergy towards latex or plastic
* Bleeding disorder

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-06-10 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Ad-libitum food intake | 120 min
  Neurotensin (NT), saline, GLP-1 and GLP-1+Neurotensin will be infused on four occasions in random order, double blinded. After 2h of infusion an ad libitum meal will be served. When the meal is completed food intake will be determined by weighing the leftovers.

SECONDARY OUTCOMES:
Appetite and gastrointestinal sensations | -60, -30, 0, 30, 60, 90, 120, 150 and 180 min
  Using visual analogue scales (VAS) the effect of infusions and meals will be documented.
  Ad libitum meals will also be evaluated using VAS.
Plasma glucose | -60, -30, 0, 15, 30, 45, 60, 90, 120, 150, 165 and 180 min
  Bed-side measurements of plasma glucose
Neurotensin | -60, -30, 0, 15, 30, 45, 60, 90, 120, 150, 165 and 180 min
  Plasma analysis
GLP-1 | -60, -30, 0, 15, 30, 45, 60, 90, 120, 150, 165 and 180 min
  Plasma analysis
Insulin | -60, -30, 0, 15, 30, 45, 60, 90, 120, 150, 165 and 180 min
  Serum analysis
C-peptide | -60, -30, 0, 15, 30, 45, 60, 90, 120, 150, 165 and 180 min
  Serum analysis
Bile acids | -60, -30, 0, 15, 30, 45, 60, 90, 120, 150, 165 and 180 min
  Plasma analysis
Ghrelin | -60, -30, 0, 15, 30, 45, 60, 90, 120, 150, 165 and 180 min
  Plasma analysis
Peptide YY (PYY) | -60, -30, 0, 15, 30, 45, 60, 90, 120, 150, 165 and 180 min
  Plasma analysis
Leptin | -60, -30, 0, 15, 30, 45, 60, 90, 120, 150, 165 and 180 min
  Plasma analysis
Metabolomics | -60, -30, 0, 15, 30, 45, 60, 90, 120, 150, 165 and 180 min
  Plasma analysis
Proteomics | -60, -30, 0, 15, 30, 45, 60, 90, 120, 150, 165 and 180 min
  Plasma analysis

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - University of Copenhagen, Department of Biomedical Scienses, Copenhagen
  - Copenhagen University Hospital Hvidovre, Copenhagen

IPD SHARING:
Plan to Share IPD: No